CLINICAL TRIAL: NCT02653950
Title: Traditional Septoplasty Vs Endoscopic Septoplasty for Treating Deviated Nasal Septum: A Prospective, Randomized Controlled Trial
Brief Title: Traditional Septoplasty Vs Endoscopic Septoplasty for Treating Deviated Nasal Septum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, SHOROOK NA'ARA MD, MD, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0576-15-RMB
Record Dates: First submitted 2016-01-06; First posted 2016-01-13 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Intranasal Surgery

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Traditional (Active Comparator): a control arm of patients undergoing traditional septoplasty for DNS
  Interventions: Procedure: Traditional septoplasty
- Endoscopic (Experimental): patients undergoing endoscopic septoplasty.
  Interventions: Procedure: Endoscopic septoplasty

INTERVENTIONS:
Procedure: Endoscopic septoplasty — Endoscopic surgery; septoplasty with or without middle turbenectomy
  Arms: Endoscopic
Procedure: Traditional septoplasty — septoplasty under direct vision
  Arms: Traditional

SUMMARY:
In this study the investigators aim to assess whether endoscopic septoplasty is effective at improving patients QOL and reducing postoperative signs and complications.

Primary outcome: To assess the differences in overall QOL between endoscopic and traditional septoplasty after adjusting for pertinent confounding variables.

Secondary outcomes:

1. To evaluate the post-operative complication rate in patients undergoing endoscopic septoplasty compared to traditional.
2. To evaluate the differences in the operation time between the two different approaches.

DETAILED DESCRIPTION:
Nasal obstruction is one of the most common complaints that the otorhinolaryngologist faces in the daily practice. Deviated nasal septum (DNS) is a very frequently encountered and common cause. It not only causes breathing difficulties but also results in improper aeration of paranasal sinuses predisiposing to sinusitis and also results in drying of mucosa leading to crusting and epistaxis 1,2. DNS can also be accompanied with hypertrophic nasal turbinates causing sleep disturbances and snoring3.

Septoplasty is an accepted and common surgical intervention to improve the nasal airway4 and sleep disturbances3.

Traditional septoplasty procedure involves sum mucosal resection of the anterior septum. The results for long-term symptom relief after traditional septoplasty are contradictory in reviewed publications 5.

In the last two decades the endoscopic Sino nasal surgery has been widely used including endoscopic approach for septoplasty. Endoscopic septoplasty as a minimally invasive technique where the dissection of the nasal septal flap can be limited minimizing trauma. The excellent visualization is presumed to decrease morbidity and post-operative swelling in isolated septal deviation by limiting the excision to the area of deviation 2. Furthermore, diagnosing and treating abnormalities of the lateral wall of the nose at the same sitting is only feasible in the endoscopic approach.

At the time of this study, there are no studies comparing the changes of quality of life in patients undergoing traditional septoplasty Vs endoscopic septoplasty.

The investigators aimed to assess whether endoscopic septoplasty is effective at improving patients QOL and reducing postoperative signs and complications.

Aims

Primary:

1) To assess the differences in overall QOL between endoscopic and traditional septoplasty after adjusting for pertinent confounding variables.

Secondary:

1. To evaluate the post-operative complication rate in patients undergoing endoscopic septoplasty compared to traditional.
2. To evaluate the differences in the operation time between the two different approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of nasal obstruction and deviated nasal septum with or without hypertrophy of nasal turbinates.
2. Patient undergoing surgery for repairing the deviated nasal septum.

Exclusion Criteria:

1. Diagnosis of bilateral acute or chronic rhinosinusitis or nasal polyposis
2. Patients undergoing endoscopic sinonasal surgery.
3. Diagnosed with inflammatory (e.g. Wegener's granulomatosis, sarcoidosis) or neoplastic nasal pathology
4. Diagnosed with systemic conditions affecting the nose e.g. Cystic fibrosis, Kartagener's syndrome
5. Patients listed for revision surgery
6. Neoplasms - untreated or under active or recent treatment with chemotherapy or radiotherapy
7. Unable to give informed consent due to mental impairment
8. Unable to adhere follow up or treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-02; Primary Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of life | Baseline (maximum 3 months before surgery), at 2-3 weeks, and 3-4 months after the surgery.
  quality of life will assessed using Sino-Nasal Outcome Test-22 (SNOT-22) scores.

REFERENCES:
- [Derived] Na'ara S, Kaptzan B, Gil Z, Ostrovsky D. Endoscopic Septoplasty Versus Traditional Septoplasty for Treating Deviated Nasal Septum: A Prospective, Randomized Controlled Trial. Ear Nose Throat J. 2021 Nov;100(9):673-678. doi: 10.1177/0145561320918982. Epub 2020 Apr 27. PMID 32339048